CLINICAL TRIAL: NCT04448834
Title: A Phase 2 Single Arm, Multicenter Trial to Evaluate the Efficacy of the BiTE® Antibody Blinatumomab (Blincyto) and Vincristine Sulfate Liposomal Injection (Marqibo) in Adult Subjects With Relapsed/Refractory Philadelphia Negative CD19+ Acute Lymphoblastic Leukemia
Brief Title: Blincyto Amgen Acrotech BioPharma PH2 Blincyto Marqibo R/R Philadelphi CD19+ ALL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not moving forward
Sponsor: Dorothy Sipkins, MD, PhD (Other)
Collaborators: Amgen (Industry); Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dorothy Sipkins, MD, PhD, Instructor in the Department of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104913
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): A single cycle of blinatumomab which includes 4 weeks of CIVI of blinatumomab followed by a 2 week treatment free interval
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — liposomal vincristine 2.25 mg/m2 weekly x 3 per cycle (weeks 3-5 in cycle 1 and 2-4 in subsequent cycles)
  Other Names: liposomal vincristine

SUMMARY:
Hypotheses: The Investigator hypothesizes that targeting ALL cells with 2 different modalities, ie liposomal vincristine sulfate as a microtubule inhibitor and blinatumomab as a BITE immuno-oncology therapy, will have at least additive benefits and allow an effective, safe therapeutic option for patients. Further, the Investigator hypothesizes that the combination will result in a high rate of response and thus allow enhanced immunologic recovery.

Primary Objectives To evaluate whether the combination will result in a median progression-free survival (PFS) of at least 1 year.

To evaluate if the complete remission/complete remission with incomplete hematological recovery (CR/CRi*) rate is ≧ 75% following 2 cycles in adult subjects with R/R Ph- ALL and duration of remission Secondary Objectives To evaluate the rate of Minimal Residual Disease (MRD) and duration To evaluate the proportion of patients who are able to progress to allogeneic transplantation To evaluate the safety of blinatumomab and liposomal vincristine sulfate in combination To evaluate the effect of the combination and response on measures of immune reconstitution

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ph-, CD19+ ALL, with any of the following:
* Relapsed or refractory to at least 2 prior regimens ≥ 5% blasts in the bone marrow or peripheral blood or persistent extranodal/marrow site (such as skin).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Age ≥ 18 years of age, at the time of informed consent.
* Subject has provided informed consent. Those unable to provide consent for themselves will not be eligible.
* Pts may have been exposed to either agent in the past if they had at least 6 months of response from start of therapy AND it has been at least 6 months since their last dose of either agent.

Exclusion Criteria:

* History of malignancy other than ALL within 3 years prior to start of protocol-required therapy with the exception of:
* Malignancy treated with curative intent and with no known active disease present for 2 years before enrollment and felt to be at low risk for recurrence by the treating physician
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease
* Adequately treated breast ductal carcinoma in situ without evidence of disease
* Prostatic cancer without evidence of progression for 1 year.
* History or presence of clinically relevant CNS pathology as adult seizures, recent stroke (within 1 year), severe brain injuries, Parkinson's disease, psychosis
* With the exception of CNS leukemia that is well controlled with therapy prior to enrolling on this study. A negative CNS evaluation for active disease is required within 3 months of enrollment in those with prior history within one year of active CNS disease .
* Current severe autoimmune disease or history of autoimmune disease with potential CNS involvement such as lupus, sjogren's, psoriasis, multiple sclerosis, wegener's granulomatosis.
* Allogeneic HSCT within 12 weeks prior to start of blinatumomab/marqibo
* Any active acute Graft-versus-Host Disease (GvHD) grade 2 to grade 4 according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment of more than 10 mg prednisone daily (or equivalent)
* Cancer chemotherapy or immunotherapy within 2 weeks prior to start of blinatumomab/marqibo. Administration of dexamethasone and hydrea permitted within the 21 day screening period.

Subject received prior anti-CD19 therapy ARE eligible however if they received prior blinatumomab, however they are ineligible if they did not have a response to it lasting at least 6 months; also they are ineligible if they had exposure to blinatumomab within 6 months of starting therapy on this study.

* Abnormal screening laboratory values as defined below:
* AST (SGOT) and/or ALT (SGPT) and/or alkaline phosphatase ≥ 5 x upper limit of normal (ULN)
* Total bilirubin ≥ 3 x ULN (unless related to Gilbert´s or Meulengracht disease)
* Creatinine ≥ 3 ULN or creatinine clearance < 40 mL/min (calculated)
* Known infection with human immunodeficiency virus (HIV) or chronic active infection with hepatitis B virus (PCR positive) or hepatitis C virus (PCR positive).
* Subject is pregnant or breast feeding
* Woman of childbearing potential and is not willing to use 2 highly effective methods of contraception while receiving blinatumomab/marqibo and for an additional 3 months after the last dose of protocol-specified therapy
* Male who has a female partner of childbearing potential, and is not willing to use 2 highly effective forms of contraception for at least an additional 3 months after the last dose of protocol-specified therapy
* Male who has a pregnant partner, and is not willing to use a condom during sexual activity for 3 months after the last dose of protocol-specified therapy
* Currently receiving treatment in another investigational device or drug study or less than 30 days since ending treatment on another investigational device or drug study(s). The 30 days is calculated from day 1 of blinatumomab treatment.
* Subject has known severe sensitivity to immunoglobulins or any of the products or components to be administered during dosing.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At 1 year
  patient report
Complete remission/complete remission with incomplete hematological recovery (CR/CRi*) rate | End of Cycle 2 (1 cycle is 6 weeks in duration)
  lab reports

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) and duration | End of Cycle 2 (1 cycle is 6 weeks in duration)
  Flow Measurement
Minimal Residual Disease (MRD) and duration | End of Therapy (up to 58 weeks)
  Flow Measurement
Proportion of patients able to progress to allogeneic transplantation | End of study (up to 58 weeks)
  Investigator reported
Safety of blinatumomab and liposomal vincristine sulfate in combination, as measured by rate of toxicity | Through all cycles of therapy (up to 58 weeks)
  Investigator report of toxicities
Immune reconstitution, as measured by the immune reconstitution panel | End of study (up to 58 weeks)
  immune reconstitution panel

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sipkins, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Duke University, Durham, North Carolina
  - Novant Health Cancer Institute and Innovation Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No